CLINICAL TRIAL: NCT04271436
Title: Early Assessment of Response to Immune Checkpoint Blockade Therapy Using 18F-FLT PET/CT
Brief Title: Immune Checkpoint Blockade Therapy Using 18F-FLT PET/CT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201909060
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET/CT + PET/MR (Experimental): -Eligible patients will have imaging assessments (as part of the study) performed at three time-points: pre-treatment, following cycle 1 of treatment, and following cycle 2 of treatment. Baseline FDG PET/CT will be a standard-of-care procedure. If possible, PET/CT imaging will be performed, followed immediately by PET/MR imaging during each imaging session. At minimum, PET/MR should be obtained at least once during each time-point (i.e. either during the FDG or FLT procedure). FDG imaging and FLT imaging should be performed at least 24 hours apart and no more than 7 days apart.
  Interventions: Device: FDG PET/CT; Device: FLT PET/CT; Device: PET/MR; Drug: [F-18] flurothymidine

INTERVENTIONS:
Device: FDG PET/CT — A single dose of 10 mCi FDG will be given by bolus injection approximately 60 minutes prior to the first planned imaging procedure.
Device: FLT PET/CT — . A single dose of 10 mCi FLT will be given by bolus injection approximately 80 minutes prior to the first planned imaging procedure.
Device: PET/MR — MR imaging will be performed on a Siemens Biograph mMR or an MRI scanner, if the PET/MR is unavailable.
Drug: [F-18] flurothymidine — -Radiopharmaceutical

SUMMARY:
In the current study, advanced positron emission tomography/computed tomography (PET/CT) and positron emission tomography/magnetic resonance (PET/MR) imaging methods will be used to validate the hypothesis that participants receiving immune checkpoint blockade (ICB) therapy, who ultimately achieve clinical benefit, will show an increase, or "FLARE", in tumor FLT and/or FDG uptake from baseline, as seen after cycle#1 of treatment, and that after 2 cycles of treatment responders will have a decline in FLT and FDG uptake, in comparison to the participants classified as "non-responders".

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of cancer.
* Patients who are planned to receive checkpoint blockade therapy, per referring oncologist.
* Life expectancy ≥ 6 months and < 5 years.
* Disease that is measurable per RECIST 1.1.
* Age ≥18 years.
* Ability and willingness to provide informed consent
* Women of child-bearing potential must have a negative urinary or serum pregnancy test within 7 days of each imaging time point.

Exclusion Criteria:

* Patient receiving other investigational radiotracers within 14 days prior to FLT and FDG imaging time points.
* Patients receiving ICB in combination with chemotherapy.
* Immunosuppressive therapy including systemic corticosteroids except for maintenance dosing for adrenal insufficiency. Patients requiring immunosuppressive therapy during the study will no longer be eligible.
* Known additional malignancy that is progressing or requires active treatment with the exceptions of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune diseases, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a pacemaker, stainless steel aneurysm clip or any other magnetic resonance (MR) contraindicated implant or foreign body would warrant exclusion from this study. Pacemakers may be reprogrammed or turned off by the strong MRI magnetic field. Radio-frequency (RF) fields in MR can also cause severe heating of pacemaker lead tips. Steel aneurysm clips are prone to torque in the strong MR field which can displace the clips and may damage the vessel, resulting in hemorrhage, and/or death.
* Pregnant women are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in FLT uptake | Between pre-treatment PET/CT imaging and end of cycle 1 PET/CT imaging (estimated to be 1 month)
  * Participants will be designated as responders or non-responders based on follow-up RECIST 1.1 measurements
  * Changes in FLT uptake will be compared between the two groups
Change in FLT uptake | Between pre-treatment PET/CT imaging and end of cycle 2 PET/CT imaging (estimated to be 2 months)
  * Participants will be designated as responders or non-responders based on follow-up RECIST 1.1 measurements
  * Changes in FLT uptake will be compared between the two groups

SECONDARY OUTCOMES:
Change in FDG uptake | Between pre-treatment PET/CT imaging and end of cycle 1 PET/CT imaging (estimated to be 1 month)
  * Participants will be designated as responders or non-responders based on follow-up RECIST 1.1 measurements
  * Changes in FDG uptake will be compared between the two groups
Change in FDG uptake | Between pre-treatment PET/CT imaging and end of cycle 2 PET/CT imaging (estimated to be 2 months)
  * Participants will be designated as responders or non-responders based on follow-up RECIST 1.1 measurements
  * Changes in FDG uptake will be compared between the two groups
Change in apparent diffusion coefficient (ADC) on diffusion-weighted MRI (DW-MRI) | From baseline to the end of second cycle of treatment (estimated to be 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wahl, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with other researchers. The researchers may be doing research at Washington University, at other research centers and institutions, or industry sponsors of research. Data may also be shared with large data repositories. The researchers may be doing research in areas similar to this research or in other unrelated areas.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 3 months and ending 10 years following article publication.
Access Criteria: Proposals should be submitted directly to rwahl@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu